CLINICAL TRIAL: NCT04513067
Title: A Phase Ib, Open-label, Dose-escalation Study of YQ23 as a Single Agent and in Combination With Pembrolizumab Administered to Patients With Advanced Solid Tumors
Brief Title: A Safety Study of YQ23 in Advanced Solid Tumors Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to business decision
Sponsor: New Beta Innovation Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YQ23-19002
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation study composed of 2 stages. Single agent in Stage 1 (as defined as arm 1) and combination therapy in Stage 2 (as defined in arm 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage 1: Single agent (Experimental): Intravenous weekly dose of YQ23 for 6 weeks with an ascending dose levels of 20, 30, 60, 90 and 120 mg/kg will be evaluated.
  Interventions: Biological: YQ23
- Stage 2: Combination Therapy (Experimental): Intravenous weekly dose of YQ23 for 6 weeks with an ascending dose levels from 20 mg/kg to the MTD obtained from Stage 1 in combination of a fixed dose of 200 mg intravenous pembrolizumab given on the same day following YQ23 administration and every 3 weeks thereafter.
  Interventions: Combination Product: Pembrolizumab

INTERVENTIONS:
Biological: YQ23 — YQ23 as a single agent will be given in Stage 1.
  Arms: Stage 1: Single agent
Combination Product: Pembrolizumab — Pembrolizumab will be given in combination with YQ23 in Stage 2
  Arms: Stage 2: Combination Therapy

SUMMARY:
This is an early phase dose escalation study which is divided into two stages: (1) Single agent of the test drug YQ23, and (2) in combination with pembrolizumab administered to patients with advanced solid tumors.

The purpose of the study is find out the safety and tolerability profile, as well as maximum tolerated dose (MTD) of YQ23 as single agent (stage 1) and in combination with pembrolizumab (stage 2). Stage 2 will start only when the MTD of single agent YQ23 has been established in Stage 1.

The distribution of YQ23 in the blood, the tumor response to YQ23 (and pembrolizumab in stage 2), the change of some pre-defined biomarkers in the tumor tissues and blood, and the change of antibody response and its relationship with the disease response, safety and drug level in the blood will also be evaluated.

In stage 1, eligible patients will be given intravenous infusion of YQ23 weekly for 6 weeks. In stage 2, eligible patients will be also be given a fixed dose of pembrolizumab 200 mg on Day 1 and every 3 weeks thereafter in addition to the weekly dose of YQ23. Dose escalation decision will be made based on the safety data available for the 6 weeks study treatment(s).

Patients may continue study treatment(s) beyond 6 weeks if s/he tolerates the study drug(s) well, the disease does not get worse after first 6 doses and meet all treatment continuation criteria, as judged by the study doctor.

DETAILED DESCRIPTION:
This is a phase 1b, open-label, dose-finding study to primarily evaluate the safety and tolerability, and MTD of YQ23 as a single agent and when in combination with pembrolizumab ("combo therapy") in patients with advanced malignant solid tumors of which it will have the potential to benefit from immunotherapy, such as triple negative breast cancer, colorectal cancer, liver cancer, non-small cell lung cancer, or renal cell carcinoma. In the study, the Pharmacokinetics (PK) profile and the disease response to YQ23 will be investigated while the Pharmacodynamics (PDx) profile and immunogenicity of YQ23 will be explored when YQ23 is given alone and in combo therapy.

The study composes of 2 stages. Stage 1 is a YQ23 alone dose escalation study; and Stage 2 is YQ23 in combination with pembrolizumab dose escalation study. The primary objective of the study is to establish the MTD of YQ23 as a single agent and the MTD when given in combination with pembrolizumab, by evaluating the incidence of dose-limiting toxicities (DLT).

In Stage 1, trial subjects will be enrolled successively in the treatment cohorts of 5 dose levels of YQ23. Each subject will receive an intravenous fixed dose of YQ23 weekly in one of the treatment cohorts. Stage 2 will start only when the MTD of single agent YQ23 has been established in Stage 1. In Stage 2, trial subjects will be enrolled successively in combo therapy dose cohorts starting with the lowest tested dose of YQ23 up to the MTD established in Stage 1. In each cohort of Stage 2, a fixed dose of 200 mg pembrolizumab will be given every 3 weeks on the same day following YQ23 administration.

Dose escalation decision will be made by an Independent Data Safety Monitoring Committee (DSMC) as determined by the DLT which is based on the incidence and intensity of drug-related adverse events (toxicities) occurring up to 5 days after the administration of the sixth dose of YQ23 in the single and combo therapy. The toxicities will be graded by the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) v5.0.

At least 3 evaluable subjects will be treated per dose cohort. Evaluable subjects are defined as subjects who have completed the first 6 doses of YQ23 and the safety assessment at Day 6 post YQ23 Dose 6, or subjects who have discontinued treatment due to a DLT. Dose escalation will only be started after all subjects in the previous cohort have completed assessments at Day 6 post Dose 6 of YQ23 in the single and combo therapy dose escalations. A satisfactory review of the safety and tolerability data by the DSMC is required before any dose escalation.

Following a 3+3 design, the MTD is defined as the highest dose level at which six patients are treated and one DLT has been observed, or three patients are treated and no one has experienced a DLT. If no DLT is found, the highest dose will be determined as the MTD.

ELIGIBILITY:
Inclusion Criteria:

* Females or males age ≥ 18 years at the time of informed consent
* Patients with histologically or cytologically confirmed solid tumors with the potential to benefit from immunotherapy, such as triple negative breast cancer, colorectal cancer, liver cancer, non-small cell lung cancer, or renal cell carcinoma, who have progressed despite prior standard therapy or are intolerant of the standard therapy, or for whom no standard therapy exists. Patients with colorectal cancer should have received prior second-line therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
* At least one measurable target lesion as outlined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria at baseline
* Must have a site of disease amenable to biopsy and not chosen as target or non-target lesions for tumor response assessment (RECIST 1.1)
* Expected life expectancy of ≥ 12 weeks
* Adequate bone marrow function at screening:

  * Hemoglobin > 8.5 g/dl
  * Absolute neutrophil count (ANC) > 1.5 x 10^9/L
  * Platelet count ≥ 75 x 10^9/L
  * PT-INR < 1.5 or APTT < 1.5 x upper limit of normal
* Adequate liver function at screening:

  * Total bilirubin ≤ 1.5 x upper limit of normal
  * Serum AST and ALT ≤ 2.5 x upper limit of normal
* Adequate renal function at screening:

  * Serum creatinine <1.5 x upper limit of normal and creatinine clearance (using Cockcroft Gault formula) > 50 mL/min
* Willing to receive bovine products
* Able to provide written informed consent
* Willing and able to comply with all aspects of the study

Exclusion Criteria:

* Subjects who have received any anti-cancer treatment or investigational agent within 21 days prior to the first dose of the trial treatment
* Any surgery or radiotherapy within 28 days prior to the first dose of the trial treatment
* Any toxic effects (except <= Grade 2: hair loss, vomiting, nausea, sensory neuropathy, endocrinopathies under stable dose of replacement therapy and abnormalities of thyroid hormones) of the prior therapy which have not been resolved to Grade 1 or less (based on CTCAE v.5.0)
* Subjects who have been discontinued from treatment due to drug-related toxicities with prior therapy directed against the same target as pembrolizumab
* Subjects who have received any anti-CTLA-4 monoclonal antibodies in the past
* Symptomatic central nervous system (CNS) metastases
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1) or any cancer curatively treated > 3 years prior to study entry
* Any history of or current active cardiac disease/dysfunction including, but not limited to, any of the following:

  1. Cardiomyopathy
  2. Congestive heart failure > NYHA class 2
  3. Coronary artery disease e.g. myocardial infarction, angina pectoris and symptomatic pericarditis
  4. Cardiac arrhythmias, e.g. supraventricular, ventricular or bradyarrhythmias
  5. 12-lead electrocardiogram parameters at screening: QTc interval > 450 msec, PR interval > 220 msec, or QRS duration > 109 msec
  6. Echocardiogram left ventricular ejection fraction < 60% as determined by echocardiography at screening
  7. Abnormal MRI cardiac perfusion scan at screening
  8. Abnormal cardiac symptoms at screening: bradycardia (heart rate < 50 beat/min at rest), tachycardia (heart rate > 90 beat/min at rest)
  9. Uncontrolled hypertension or a supine systolic blood pressure > 160 or < 90 mmHg at screening
* Known connective tissue disease
* Active or known autoimmune disease. (Note: Patient with vitiligo, type I diabetes mellitus, residual hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll)
* Active or known hemolytic disorder
* Subjects receiving chronic treatment with systemic (oral/intravenous) steroid therapy (> 10mg/day prednisone or equivalent) within 7 days prior to the first dose of trial treatment.
* Subjects receiving chronic treatment with systemic (oral/intravenous) immunosuppressive medication that may interfere with the action of the trial treatment
* Known to be serologically positive for human immunodeficiency viruses (HIV)
* Patients with active Hepatitis B infection (HBsAg positive) and not adequately controlled by antiviral with HBV DNA >1000 IU/mL shall be excluded
* Patients with a positive test for hepatitis C ribonucleic acid
* Co-existing active infection requiring parenteral antibiotics or serious concurrent illness deemed clinically significant within 4 weeks prior to the first dosing of the study drug.
* Patients with a seizure disorder requiring medication (such as steroids or anti-epileptics)
* Patients undergoing renal dialysis
* Patients with clinically significant proteinuria at screening (clinically significant proteinuria is defined as urinary protein >=3.5g/24 hours)
* Patients who have received organ transplantation
* Patients who have received blood transfusion within 4 weeks prior to trial treatment
* Known hypersensitivity to any blood product and therapeutic antibody
* Known allergy to bovine products
* Patients who have received bovine hemoglobin-based oxygen carrier (HBOC) or other HBOC in the past
* Female who is pregnant or breast-feeding at screening or baseline
* Female of childbearing potential who is not willing to use 2 methods (1 primary and 1 secondary method) of birth control throughout the trial treatment period and for 6 months after discontinuation of the treatment
* Male subject with female partner of childbearing potential is not willing to use a male barrier method of contraception (i.e. male condom with spermicide) in addition to a second acceptable contraception method throughout the treatment period and for 6 months after discontinuation of the treatment
* Any condition that is unstable or could jeopardize the safety of the subjects and their compliance in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) of YQ23 as single agent (Stage 1) and when in combination with Pembrolizumab (Stage 2) | From start of study until 12 weeks after last dose
  The incidence and severity of AEs and SAEs including the following cardiac events of interests evaluated by Common Terminology Criteria for Adverse Events (CTCAE) v5.0:
  * High-sensitivity cardiac troponin I increase
  * Ejection fraction decrease
  * Electrocardiogram corrected QT interval prolongation
  * Creatine phosphokinase increase
Establishment of MTD for YQ23 as single agent (Stage 1) and when in combination with Pembrolizumab (Stage 2) | From the start of treatment until Day 6 post Dose 6 of YQ23 at each dose level (in both stages)
  MTD will be evaluated by the incidence of DLT for which it will be determined based on the incidence and intensity of drug-related adverse events (toxicities) occurring up to 8 days after the administration of the fourth dose of YQ23 in the single and combo therapy dose escalations. The toxicities will be graded by the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Pharmacokinetics of YQ23 as measured by plasma concentration in single agent group and combo therapy group | Pre-dose, 0hour (End of infusion, EoI), 0.25hour, 0.5hour, 1hour, 2hours, 6hours, 12hours, 24hours, 48hours post-EoI of the initial dose and 0.5hour post-EoI Dose 6
  Plasma level of YQ23 will be serially evaluated following dosing of study drug(s), and the maximum observed plasma concentration (Cmax) of YQ23 will be determined.
Pharmacokinetics of YQ23 as measured by area under the plasma concentration-time curve in single agent group and combo therapy group | Pre-dose, 0hour (End of infusion, EoI), 0.25hour, 0.5hour, 1hour, 2hours, 6hours, 12hours, 24hours, 48hours post-EoI of the initial dose and 0.5hour post-EoI Dose 6
  Plasma level of YQ23 will be serially evaluated following dosing of study drug(s), and area under the plasma concentration-time curve of YQ23 will be determined.
Pharmacokinetics of YQ23 as measured by terminal half-life in single agent group and combo therapy group | Pre-dose, 0hour (End of infusion, EoI), 0.25hour, 0.5hour, 1hour, 2hours, 6hours, 12hours, 24hours, 48hours post-EoI of the initial dose and 0.5hour post-EoI Dose 6
  Plasma level of YQ23 will be serially evaluated following dosing of study drug(s), and terminal half-life of YQ23 will be determined.
Disease control rate (DCR) by YQ23 when given alone and when in combination with pembrolizumab | This will be measured at Day 6 post YQ23 Dose6
  DCR is defined as the proportion of patients with the best overall response of complete response (CR) or partial response (PR) or stable disease (SD) using RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Billy Lau, PhD., Study Director — New Beta Innovation Limited
Locations (1):
- The University of Hong Kong Phase I Clinical Trials Centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No